CLINICAL TRIAL: NCT03201380
Title: Evaluation of the Practice of the TEP Choline in Provence - Alps and Côte d'Azur at Patients With Prostate Cancer - Multicentre Retrospective Study.
Brief Title: Evaluation of the Practice of the TEP Choline at Patients With Prostate Cancer
Acronym: TEPCholine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: TEP Choline-IPC 2016-007
Record Dates: First submitted 2017-06-16; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Choline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TEP scanner with choline

SUMMARY:
The prostate cancer is a heterogeneous disease the care of which varies according to the status: localized, locally advanced, or in recurrence after local or metastatic treatment. The precise evaluation of the degree of extension of the disease is thus essential because it is going to allow to adapt at best the therapeutic strategy.

Contrary to the abdomino-pelvic scanning and to the osseous scintigraphy which(who) are a member(part) of the balance assessment of standard extension of the prostate cancer, the place of the Tomography with broadcast of Positrons to scan (TEP scan) in Choline in the management of patients affected by prostate cancer is not clearly defined in the national and European recommendations.

The current marketing authorization ( AMM) is the research for bones localizations in the prostatic cancers at high risk. It indeed seems that this examination is more successful than the standard radiological examinations (bone scintigraphy and abdomino-pelvic scanning) in the detection of the bone metastatic hurts, with a sensibility of about 100 % and a precision of the order of 93 % according to certain studies.

The recent data of the literature suggest a quite particular interest at the patients in situation of biochemical recurrence in terms of localization of (or) tumoral site (s).

THE AMM however not specifying if this examination has to be made within the framework of the initial balance sheet of extension, at the time of the biochemical second offense or at the known metastatic stage, there is a big variability of the practices according to the centers.

The current indications being very ill-assorted, he is interesting being able to estimate the heterogeneousness of the practices of way multicentre, by leading a study observationally retrospective in region Provence-Alpes-Côte d'Azur (PACA).

ELIGIBILITY:
Inclusion Criteria:

* Have had a TEP scan in the choline
* Prostate cancer

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients having had a TEP in the choline for a prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of TEP scan in Choline indications in the care of prostate cancers and more particularly the search for bone metastasis at diagnosis | One year
  Disease evaluation method by scanner with choline
Number of TEP scan in Choline indications in the care of prostate cancers and more particularly the search for bone metastasis at the site of relapse after local treatment | One year
  Disease evaluation method by scanner with choline
Number of TEP scan in Choline indications of TEP scan in Choline in the care of prostate cancers and more particularly the search for bone metastasis during the follow-up of the disease | One year
  Disease evaluation method by scanner with choline

SECONDARY OUTCOMES:
Modifications of therapeutic strategy in the care of prostate cancers | One year
  Disease evaluation method by scanner with choline

CONTACTS AND LOCATIONS:
Overall Officials: PIGNOT Géraldine, MD, Principal Investigator — Institut Paoli-Calmettes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr